CLINICAL TRIAL: NCT06054542
Title: Validity and Reliability of the Turkish Version of Digital Eye Strain Questionnaire (DESQ)
Brief Title: Turkish Version of Digital Eye Strain Questionnaire (DESQ)
Status: Recruiting | Type: Observational
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayse Unal, Assoc. Prof., Alanya Alaaddin Keykubat University
Other Study IDs: 20.09.2023/DESQ
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cultural Adaptation; Reliability; Validity; Adults; Eye Strain
MeSH Terms: conditions — Asthenopia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cultural adaptation, reliability and validity — Cross-cultural Adaptation, Reliability and Validity of the Turkish Version of the DESQ

SUMMARY:
The aims of this study were to perform cultural adaptation of the DESQ and provide information regarding the factor structure, reliability and validity of the instrument in Turkish speaking adults.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65 years
* People who spend two or more continuous hours a day on their digital devices (computer, tablet, smartphone) or use more than one device

Exclusion Criteria:

* History of ophthalmic surgery or active ocular disease
* Participants who did not understand the instructions or did not sign a consent form were excluded

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults who spend two or more continuous hours a day on their digital devices (computer, tablet, smartphone) or use more than one device
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
DESQ | Baseline and after 7 days
  Digital Eye Strain Questionnaire (DESQ) is a thirteen-item self-report scale in a yes-no format designed to offer a measure of complaints related to digital eye strain syndrome (DES)

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Alaadin Keykubat University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No